CLINICAL TRIAL: NCT06210984
Title: The Effects of Caffeine Supplementation on Training Intensity Quantification
Brief Title: Caffeine and Training Intensity Quantification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Stmarys1
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low caffeine dose (Experimental): 2 mg/kg dose of caffeine (in pill form)
  Interventions: Drug: Low caffeine dose
- Moderate caffeine dose (Experimental): 5 mg/kg dose of caffeine (in pill form)
  Interventions: Drug: Moderate caffeine dose
- Placebo (Placebo Comparator): 5 mg/kg dose of placebo (Maltodextrin in pill form)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low caffeine dose — 2 mg/kg dose of caffeine in pill form
  Arms: Low caffeine dose
Drug: Moderate caffeine dose — 5 mg/kg dose of caffeine in pill form
  Arms: Moderate caffeine dose
Drug: Placebo — 5 mg/kg dose of maltodextrin in pill form
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the effects of caffeine on exercise physiology and the subsequent quantification of athlete training zones in trained cyclists. The main questions that it aims to answer are:

* What are the effects of low and moderate doses of caffeine on exercise physiology.
* How do the effects of caffeine on exercise physiology affect the calculation of training zones.
* Do the effects of caffeine on exercise physiology differ between men and women.

Participants will complete four trials on a cycle ergometer as follows:

* Trial 1: participants will complete two incremental tests to determine the power outputs required to elicit 50-80% of maximal oxygen consumption for trials 2-4.
* Trials 2-4: participants will consume (in a randomized order) either a low (2 mg/kg) dose of caffeine, a moderate (5 mg/kg) dose of caffeine, or a placebo (maltodextrin), 45 minutes prior to to completing an incremental cycling test from 50-80% of maximal oxygen uptake.

Measures of heart rate, oxygen uptake, blood lactate, and perceived exertion will be recorded throughout all trials.

Researchers will compare the effects of exercise intensity, caffeine dose, and sex to see if they affect exercise physiology and training zone quantification.

ELIGIBILITY:
Inclusion Criteria:

* To be considered for inclusion in the study, participants must be regular cyclists, between 18 and 45 years of age, capable of completing a 20 km cycling time trial at a minimum speed of 30 km/h for men and 28 km/h for women (arbitrary inclusion criteria to ensure a sufficient standard of athlete). Female participants must have a regular menstrual cycle and not be taking oral contraceptives.

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood lactate concentration | From baseline to completion, up to 31 days
  Change from baseline in blood lactate concentration measured at rest and at seven different exercise intensities (50, 55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer
Heart rate | From baseline to completion, up to 31 days
  Change from baseline in heart rate measured at rest and at seven different exercise intensities (50, 55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer
Oxygen uptake | From baseline to completion, up to 31 days
  Change from baseline in oxygen uptake measured at rest and at seven different exercise intensities (50, 55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer
Perceived exertion | From baseline to completion, up to 31 days
  Change from baseline in rating of perceived exertion measured (using the 6-20 Borg scale) at seven different exercise intensities (50, 55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer